CLINICAL TRIAL: NCT05590806
Title: The Effect of Ground and Unground Enamel on the Clinical Performance of Direct Composite Build-ups After Orthodontic Treatment: Five Years of Follow-up
Brief Title: The Effect of Ground and Unground Enamel on the Clinical Performance of Direct Composite Build-ups
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Demirci, Istanbul University, Istanbul University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: 2011-97
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Trial of Labor; Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Restoration
  Interventions: Other: Direct composite build-ups
- Arm 2 (Experimental): Evaluate
  Interventions: Other: Direct composite build-ups

INTERVENTIONS:
Other: Direct composite build-ups — Direct composite build-ups application

SUMMARY:
Twenty-four patients participated in the study. Patients received direct composite build-ups for diastema closure.

DETAILED DESCRIPTION:
The restorations were performed separately by grounding and ungrounding the enamel on the proximal surfaces in symmetrical teeth.

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene, no periodontal or pulpal disease, interarch tooth size discrepancies (Bolton discrepancy) after orthodontic treatment

Exclusion Criteria:

* uncontrollable parafunctions, insufficient or poor oral hygiene, periodontal or gingival disease

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Success rate | 5 years

IPD SHARING:
Plan to Share IPD: No